CLINICAL TRIAL: NCT04266366
Title: Comparison of Cost and Cost- Effectiveness of a Face-to-Face Rehabilitation Program vs an Telemedicine Program on Disability, Pain, Fear of Movement, Quality of Life and Spinal Mobility in Patients With Chronic Low Back Pain
Brief Title: Cost- Effectiveness of a Face-to-Face Rehabilitation Program vs an Telemedicine Program in Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Collaborators: Junta de Andalucia (Other Government)
Responsible Party: Principal Investigator, Adelaida María Castro-Sánchez, Principal Investigator, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CE-IP00562
Record Dates: First submitted 2020-02-07; First posted 2020-02-12 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Low Back Pain
Keywords: Low back pain; Electroanalgesia; McKenzie Method; Telemedicine; Study protocol for a Randomized clinical trial
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Study protocol for a double blinded two-arm randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Face-to Face rehabilitation program (Active Comparator): Electroanalgesia therapy and the McKenzie exercise protocol will be applied by six therapists with more than 10 years of experience. This program will be developed in the rehabilitation service of the study health centers. Patients will perform the treatment 3 times per week, for 4 weeks, with a total of 24 sessions
  Interventions: Other: Face-to-Face Rehabilitation program
- Telemedicine Program (Experimental): It consists in a support system for the treatment of chronic low back pain based on web technologies. The system can register a subject and provide a treatment of electroanalgesia and exercise through the Mckenzie method. Video applications of electroanalgesia and exercises will be shown to patients who use their computer or mobile device to access the platform through the Internet. The treatments will be recommended by the system based on the database that is configured to accommodate the application of electroanalgesia and McKenzie exercises based on the diagnosis according to the McKenzie method.patients will perform the treatment 3 times per week, for 8 weeks, with a total of 24 sessions
  Interventions: Other: Telemedicine program

INTERVENTIONS:
Other: Face-to-Face Rehabilitation program — In each hospital, two trained therapists will carry out a face-to-face rehabilitation program consisting of electroanalgesia and an exercise program that follows the Mckenzie method. The physiotherapists place the electrodes in the patients, for this they use 5x9 cm electrodes, which they place at the bilateral paravertebral level, in the patients who present with radicular pain, the electrodes will be placed in the path of the affected nerve. The duration will be sufficient to carry out the Mckenzie protocol. Mckenzie exercises are designed to make changes in the internal periarticular components of the spine.
  Arms: Face-to Face rehabilitation program
Other: Telemedicine program — It consists in an e-Health rehabilitation program through a web platform performing electroanalgesia and an exercise program following the Mckenzie method. Patients will be instructed in the use of the TENS device using 5x9cm electrodes at the bilateral paravertebral level, the patients that present radicular pain, the electrodes will be placed in the path of the affected nerve. The realization of exercises will be through the application of an Mckezie protocol. The duration will be the same as that used to carry out the Mckenzie protocol. Mckenzie exercises are designed to make changes in the internal components periarticular of the spine.
  Arms: Telemedicine Program

SUMMARY:
Perform a cost-utility analysis in patients with chronic low back pain through electroanalgesia treatment and exercises administered by telemedicine program versus face-to-face program

DETAILED DESCRIPTION:
A double blind clinical trial will be developed in a sample of 80 subjects with chronic low back pain. Patients will receive 3 weekly sessions of electroanalgesia and an exercise program for 8 weeks, for a total of 24 sessions. The aim is to analyze the cost- effectiveness of a face-to- face rehabilitation program vs a telemedicine program on disability, pain, fear of movement, quality of life, resistance of the trunk flexors, lumbar mobility in flexion and muscular electrical activity.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain ≥ 3 months.
* Age between 30 and 67 years old.
* Not being receiving physical therapy.

Exclusion Criteria:

* Presence of lumbar stenosis.
* Diagnosis of spondylolisthesis.
* Diagnosis of fibromyalgia.
* Treatment with corticosteroids or oral medication in recent weeks.
* History of spine surgery.
* Contraindication of analgesic electrical therapy.
* Have previously received a treatment of electrical analgesia or exercise.
* Central or peripheral nervous system disease.

Ages: 30 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Roland Morris Disability Questionnaire (RMDQ). | At baseline, at 8 weeks and at 6 months
  This is a self-reported questionnaire consisting in 24 items reflecting limitations in different activities of daily living attributed to low back pain including walking, vending over, sitting, lying down, dressing, sleeping, self-care and daily activities.Ranging from 0 points- better to 24 points- worse disability

SECONDARY OUTCOMES:
Change from baseline in disability. Oswestry Low Back Pain Disability Idex. | At baseline, at 8 weeks and at 6 months.
  It has 10 items associated to activities of daily living, each ítem has a puntuation fron 0 to 5 points.The higher scores mean a worse outcome.
Change from baseline in pain intensity. Visual analogue scale. | At baseline, at 8 weeks and at 6 months
  A 10-point Numerical Pain Scale (0: no pain, 10: maximum pain) assesses the intensity of pain. Range from no pain 0 to maximum pain 10 points
Change from baseline in Fear of Movement. Tampa Scale of kinesiophobia. | At baseline, at 8 weeks and at 6 months
  Is a 17-item questionnaire that measures the fear of movement and (re)injury.Patient rate beliefs about their kinesiophobia on a 4-point scale ranging from strongly disagree to strongly agree.
Change from baseline on Quality of Life. SF-36 Health questionnaire. | At baseline, at 8 weeks and at 6 months
  SF-36 Health questionnaire scores range from 0 to 100% and indicate the self-perceived health-related quality of life.
Change from Mcquade Test | At baseline, at 8 weeks and at 6 months
  It measures the isometric endurance of trunk flexion muscles.
Change from baseline in lumbar mobility flexion. | At baseline, at 8 weeks and at 6 months
  For the quantification of lumbar flexion an angular inclinometer is used (Fleximeter UM 8320-3 RJ Code Research Institute, Brazil).
Changes from baseline in Lumbar electromyography. | At baseline, at 8 weeks and at 6 months
  The degree of electromyographic activation of the lumbar paravertebral musculature will be carried out by using a set of electrodes of 3x7 dimensions that will be applied uniformly in the lumbar region from the spinal level from L2 to L5.
Change from baselina in range of motion | At baseline, at 8 weeks and at 6 months
  This variable is quantified using the SpinalMouse ® device (Phisiotech, Spain). It is an electronic computer-aided measuring device that measures sagittal spinal amplitude of movement (ROM) and intersegmental angles in a non-invasive way.
Change from baselina in lumbar segmental mobility | At baseline, at 8 weeks and at 6 months
  This variable is quantified using the SpinalMouse ® device (Phisiotech, Spain). It is an electronic computer-aided measuring device that measures sagittal spinal amplitude of movement (ROM) and intersegmental angles in a non-invasive way.
Change from baseline in indirect non-medical costs | At baseline, at 8 weeks and at 6 months
  sick leave days due to low back pain and labor absenteeism costs in terms of workdays lost due to illness at salary level.
Change from baseline in direct medical costs | At baseline, at 8 weeks and at 6 months
  costs of visits to primary care, emergency visits, home help received as a result of disability related to LBP, diagnostic tests and pharmaceutical products
Change from baseline direct non-medical costs | At baseline, at 8 weeks and at 6 months
  The patient expenses in transportation

CONTACTS AND LOCATIONS:
Overall Officials: Adelaida María Castro-Sánchez, PhD, Principal Investigator — Almería University
Locations (1):
- Universidad de Almería, Almería, Andalusia, Spain

REFERENCES:
- [Background] Von Korff M, Moore JC. Stepped care for back pain: activating approaches for primary care. Ann Intern Med. 2001 May 1;134(9 Pt 2):911-7. doi: 10.7326/0003-4819-134-9_part_2-200105011-00016. PMID 11346328
- [Background] Schaafsma FG, Whelan K, van der Beek AJ, van der Es-Lambeek LC, Ojajarvi A, Verbeek JH. Physical conditioning as part of a return to work strategy to reduce sickness absence for workers with back pain. Cochrane Database Syst Rev. 2013 Aug 30;2013(8):CD001822. doi: 10.1002/14651858.CD001822.pub3. PMID 23990391
- [Background] Becker A, Held H, Redaelli M, Strauch K, Chenot JF, Leonhardt C, Keller S, Baum E, Pfingsten M, Hildebrandt J, Basler HD, Kochen MM, Donner-Banzhoff N. Low back pain in primary care: costs of care and prediction of future health care utilization. Spine (Phila Pa 1976). 2010 Aug 15;35(18):1714-20. doi: 10.1097/brs.0b013e3181cd656f. PMID 21374895
- [Background] Dagenais S, Caro J, Haldeman S. A systematic review of low back pain cost of illness studies in the United States and internationally. Spine J. 2008 Jan-Feb;8(1):8-20. doi: 10.1016/j.spinee.2007.10.005. PMID 18164449
- [Background] GBD 2015 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 310 diseases and injuries, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1545-1602. doi: 10.1016/S0140-6736(16)31678-6. PMID 27733282
- [Background] Froud R, Patterson S, Eldridge S, Seale C, Pincus T, Rajendran D, Fossum C, Underwood M. A systematic review and meta-synthesis of the impact of low back pain on people's lives. BMC Musculoskelet Disord. 2014 Feb 21;15:50. doi: 10.1186/1471-2474-15-50. PMID 24559519
- [Background] Palacin-Marin F, Esteban-Moreno B, Olea N, Herrera-Viedma E, Arroyo-Morales M. Agreement between telerehabilitation and face-to-face clinical outcome assessments for low back pain in primary care. Spine (Phila Pa 1976). 2013 May 15;38(11):947-52. doi: 10.1097/BRS.0b013e318281a36c. PMID 23238489
- [Background] Airaksinen O, Brox JI, Cedraschi C, Hildebrandt J, Klaber-Moffett J, Kovacs F, Mannion AF, Reis S, Staal JB, Ursin H, Zanoli G; COST B13 Working Group on Guidelines for Chronic Low Back Pain. Chapter 4. European guidelines for the management of chronic nonspecific low back pain. Eur Spine J. 2006 Mar;15 Suppl 2(Suppl 2):S192-300. doi: 10.1007/s00586-006-1072-1. No abstract available. PMID 16550448
- [Background] Jensen CE, Riis A, Petersen KD, Jensen MB, Pedersen KM. Economic evaluation of an implementation strategy for the management of low back pain in general practice. Pain. 2017 May;158(5):891-899. doi: 10.1097/j.pain.0000000000000851. PMID 28114182
- [Background] Petersen T, Kryger P, Ekdahl C, Olsen S, Jacobsen S. The effect of McKenzie therapy as compared with that of intensive strengthening training for the treatment of patients with subacute or chronic low back pain: A randomized controlled trial. Spine (Phila Pa 1976). 2002 Aug 15;27(16):1702-9. doi: 10.1097/00007632-200208150-00004. PMID 12195058
- [Background] Khadilkar A, Milne S, Brosseau L, Robinson V, Saginur M, Shea B, Tugwell P, Wells G. Transcutaneous electrical nerve stimulation (TENS) for chronic low-back pain. Cochrane Database Syst Rev. 2005 Jul 20;(3):CD003008. doi: 10.1002/14651858.CD003008.pub2. PMID 16034883
- [Derived] Castro-Sanchez AM, Mataran-Penarrocha GA, Gomez-Garcia S, Garcia-Lopez H, Andronis L, Albornoz-Cabello M, Lara Palomo IC. Study protocol randomised controlled trial comparison of cost-utility and cost-effectiveness of a face-to-face rehabilitation programme versus a telemedicine programme in the treatment of patients with chronic low back pain. BMJ Open. 2020 Dec 12;10(12):e040633. doi: 10.1136/bmjopen-2020-040633. PMID 33310802